CLINICAL TRIAL: NCT02783573
Title: A Randomized, Double-Blind, Placebo-Controlled and Delayed-Start Study of LY3314814 in Mild Alzheimer's Disease Dementia
Brief Title: A Study of Lanabecestat (LY3314814) in Participants With Mild Alzheimer's Disease Dementia
Acronym: DAYBREAK-ALZ
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: An independent assessment concluded the trial was not likely to meet the primary endpoint upon completion and therefore, trial stopped for futility.
Sponsor: AstraZeneca (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 16024; I8D-MC-AZET (Other: Eli Lilly and Company); 2015-005625-39 (EudraCT Number)
Record Dates: First submitted 2016-05-24; First posted 2016-05-26 (Estimated); Results first posted 2019-08-06 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-10

CONDITIONS: Alzheimer's Disease
Keywords: dementia; brain diseases; neurodegenerative diseases; central nervous system diseases; nervous system diseases; mental disorders; delirium, dementia, amnestic, cognitive; tauopathies; memory; amyloid
MeSH Terms: conditions — Alzheimer Disease; Dementia; Brain Diseases; Neurodegenerative Diseases; Central Nervous System Diseases; Nervous System Diseases; Mental Disorders; Delirium; Tauopathies | interventions — lanabecestat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Lanabecestat 20 milligrams (mg) (Experimental): Participants received Lanabecestat 20 mg film-coated tablets orally once daily until week 156.
  Interventions: Drug: Lanabecestat
- Lanabecestat 50 mg (Experimental): Participants received Lanabecestat 50 mg film-coated tablets orally once daily until week 156.
  Interventions: Drug: Lanabecestat
- Placebo/ Lanabecestat 20 mg (Experimental): Placebo given orally once daily for 78 weeks and then 20 mg of lanabecestat given orally once daily until week 156.
  Interventions: Drug: Lanabecestat; Drug: Placebo
- Placebo/ Lanabecestat 50 mg (Experimental): Placebo given orally once daily for 78 weeks and then 50 mg of lanabecestat given orally once daily until week 156.
  Interventions: Drug: Lanabecestat; Drug: Placebo

INTERVENTIONS:
Drug: Lanabecestat — Administered orally
  Other Names: LY3314814; AZD3293
Drug: Placebo — Administered orally
  Arms: Placebo/ Lanabecestat 20 mg; Placebo/ Lanabecestat 50 mg

SUMMARY:
The main purpose of this study is to evaluate the efficacy of the study drug known as lanabecestat in participants with mild Alzheimer's disease (AD) dementia.

ELIGIBILITY:
Inclusion Criteria:

* Participant must meet the National Institute on Aging (NIA) and the Alzheimer's Association (AA) (NIA-AA) criteria for probable AD dementia.
* MMSE score of 20 to 26 inclusive at screening visit.
* For a diagnosis of mild AD dementia, participant must have a CDR global score of 0.5 or 1, with the memory box score ≥0.5 at screening.
* Evidence of amyloid pathology.
* The participant must have a reliable study partner with whom he/she cohabits or has regular contact.

Exclusion Criteria:

* Significant and/or current neurological disease affecting the central nervous system, other than AD, that may affect cognition or ability to complete the study, including but not limited to, other dementias, repetitive head trauma, serious infection of the brain, Parkinson's disease, epilepsy, or cervicocranial vascular disease.
* Participants with any current primary psychiatric diagnosis other than AD if, in the judgment of the investigator, the psychiatric disorder or symptom is likely to confound interpretation of drug effect, affect cognitive assessment, or affect the participant's ability to complete the study. Participants with history of schizophrenia or other chronic psychosis are excluded.
* Within 1 year before the screening visit or between screening and randomization, any of the following: myocardial infarction; moderate or severe congestive heart failure, New York Heart Association class III or IV; hospitalization for, or symptoms of, unstable angina; syncope due to orthostatic hypotension or unexplained syncope; known significant structural heart disease (such as, significant valvular disease, hypertrophic cardiomyopathy); or hospitalization for arrhythmia.
* Congenital QT prolongation.
* Intermittent second- or third-degree atrioventricular (AV) heart block or AV dissociation or history of ventricular tachycardia.
* A corrected QT (QTcF) interval measurement >470 milliseconds (men and women) at screening (as determined at the investigational site).
* History of malignant cancer within the last 5 years.
* History of vitiligo and/or current evidence of post-inflammatory hypopigmentation.
* Calculated creatinine clearance <30 milliliters per minute (Cockcroft-Gault formula; Cockcroft and Gault 1976) at screening.
* Currently enrolled in any other clinical trial involving an investigational product or any other type of medical research judged not to be scientifically or medically compatible with this study.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1722 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2018-09-28 (Actual); Study Completion 2018-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (262):
- United States (90):
  - Xenoscience, Phoenix, Arizona
  - St Josephs Hospital and Medical Center, Phoenix, Arizona
  - Four Peaks Neurology, Scottsdale, Arizona
  - Arizona Neurology, Scottsdale, Arizona
  - Center for Neurosciences, Tucson, Arizona
  - NEA Baptist Clinical, Jonesboro, Arkansas
  - The Research Center of Southern California, Carlsbad, California
  - WCCT Global, Costa Mesa, California
  - Neuro-Pain Medical Center, Fresno, California
  - Neurology Center of North Orange County, Fullerton, California
  - Pacific Neuroscience Medical Group, Oxnard, California
  - California Research Foundation, San Diego, California
  - Pacific Research Network Inc, San Diego, California
  - Sharp Mesa Vista Hospital, San Diego, California
  - Syrentis Clinical Research, Santa Ana, California
  - Care Access Research, Santa Clarita, California
  - California Neuroscience Research, Sherman Oaks, California
  - Care Access Research, Valencia, California
  - Associated Neurologists, PC - Danbury, Danbury, Connecticut
  - Institute for Neurodegenerative Disorders, New Haven, Connecticut
  - Yale University School of Medicine, New Haven, Connecticut
  - Research Center for Clinical Studies, Inc, Norwalk, Connecticut
  - JEM Research Institute, Atlantis, Florida
  - Morton Plant Hospital, Clearwater, Florida
  - Brain Matters Research, Delray Beach, Florida
  - Cohen Medical Associates P.A., Delray Beach, Florida
  - Neuropsychiatric Research Center of Southwest Florida, Fort Myers, Florida
  - Indago Research & Health Center, Inc., Hialeah, Florida
  - Infinity Clinical Research, LLC, Hollywood, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Mayo Clinic-Jacksonville, Jacksonville, Florida
  - Gregory A. Kirk MD LLC, Merritt Island, Florida
  - University of Miami, Miami, Florida
  - Allied Biomedical Research Institute, Inc., Miami, Florida
  - Compass Research, Orlando, Florida
  - Quantum Laboratories, Pompano Beach, Florida
  - Charlotte Neurological Services, Port Charlotte, Florida
  - Intercoastal Medical Group, Sarasota, Florida
  - Axiom Research, Tampa, Florida
  - University of South Florida, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Atlanta Center of Medical Research, Atlanta, Georgia
  - Georgia Regents University, Augusta, Georgia
  - Medical Research Health and Education Foundation, Inc, Columbus, Georgia
  - Hawaii Medical Center, Honolulu, Hawaii
  - Advanced Clinical Research LLC, Meridian, Idaho
  - American Health Network, Avon, Indiana
  - Josephson Wallack Munshower Neurology, Indianapolis, Indiana
  - American Health Network, Muncie, Indiana
  - University of Kansas Hospital, Fairway, Kansas
  - Cotton O'Neil Clinic, Topeka, Kansas
  - Via Christi Research, Inc., Wichita, Kansas
  - Baptist Health Medical Group, Lexington, Kentucky
  - Associates in Neurology, PSC, Lexington, Kentucky
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Neurology, Scarborough, Maine
  - Boston University Medical Center, Boston, Massachusetts
  - Donald S Marks, Plymouth, Massachusetts
  - Alzheimers Disease Center, Winchester, Massachusetts
  - Michigan State University, East Lansing, Michigan
  - Hattiesburg Clinic, Hattiesburg, Mississippi
  - Clinical Research Professionals, St Louis, Missouri
  - Las Vegas Medical Research, Las Vegas, Nevada
  - Advanced Memory Research Institute of New Jersey, Toms River, New Jersey
  - Neurology Specialists of Monmouth County, West Long Branch, New Jersey
  - New York University Medical Center, New York, New York
  - Behavioral Health Center Research, Charlotte, North Carolina
  - Raleigh Neurology Associates, Raleigh, North Carolina
  - PMG Research of Winston-Salem, LLC, Winston-Salem, North Carolina
  - Wake Forest Baptist Univ CAR, Winston-Salem, North Carolina
  - Rapid Medical Research Inc, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - Insight Clinical Trials, Shaker Heights, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Cutting Edge Research Group, Oklahoma City, Oklahoma
  - The Corvallis Clinic P.C., Corvallis, Oregon
  - Summit Research Network Inc, Portland, Oregon
  - Clinical Trial Center, LLC, Psychiatry, Jenkintown, Pennsylvania
  - Pearl Clinical Research Inc., Norristown, Pennsylvania
  - Rhode Island Mood & Memory Research Institute, East Providence, Rhode Island
  - Rhode Island Hospital, Providence, Rhode Island
  - Butler Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Radiant Research, Greer, South Carolina
  - Coastal Neurology PA, Port Royal, South Carolina
  - Holston Medical Group Clinical Research, Kingsport, Tennessee
  - Univ of North Texas Health Science Center, Fort Worth, Texas
  - Texas Medical Research Associates, L.L.C., San Antonio, Texas
  - Ericksen Research and Development, Clinton, Utah
  - SSM Health Dean Medical Group, Madison, Wisconsin
- Canada (11):
  - University of Calgary, Calgary, Alberta
  - The Medical Arts Health Research Group, West Vancouver, British Columbia
  - True North Clinical Research Halifax, LLC, Halifax, Nova Scotia
  - Bruyere Continuing Care, Ottawa, Ontario
  - Kawartha Regional Memory Clinic, Peterborough, Ontario
  - Toronto Memory Program, Toronto, Ontario
  - Toronto Sunnybrook Regional Cancer Center, Toronto, Ontario
  - CSSS-Institut Universitaire Gériatric de Sherbrooke, Sherbrooke, Qubec
  - Recherches Neuro-Hippocampe Inc, Gatineau, Quebec
  - Q&T Research Sherbrooke Inc, Sherbrooke, Quebec
  - Douglas Hospital and Research Centre, Verdun, Quebec
- China (13):
  - Xuanwu Hospital-Capital Medical University, Beijing, Beijing Municipality
  - Beijing 301 Hospital, Beijing, Beijing Municipality
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - Tangshan Worker Hospital, Tangshan, Hebei
  - Nanjing Drum Tower Hosp Affiliated Hosp of Nanjing Univ Med, Nanjing, Jiangsu
  - Zhongda Hospital-Southeast University, Nanjing, Jiangsu
  - Northern Jiangsu People's Hospital, Yangzhou, Jiangsu
  - Qingdao Municipal Hospital, Qingdao, Shandong
  - Shanghai Tongji Hospital(CCBR site), Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - The First Affiliated Hospital, Zhejiang University, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical College, Wenzhou, Zhejiang
  - Shanghai Huashan Hospital Affil to Fu Dan University, Shanghai
- Czechia (9):
  - Fakultni nemocnice u sv. Anny v Brne, Brno
  - Neurohk s.r.o., Choceň
  - Neuropsychiatrie s.r.o, Hradec Králové
  - Brain-Soultherapy s.r.o, Kladno
  - A-Shine s.r.o., Pilsen
  - Clintrial, s.r.o., Prague
  - Neuropsychiatrie s.r.o, Prague
  - Medical Services Prague s.r.o., Prague
  - Axon Clinical, s.r.o., Prague
- Denmark (4):
  - CCBR-Alborg-DK, Aalborg
  - Center For Clinical and Basic Research, Ballerup Municipality
  - Rigshospitalet, Copenhagen
  - Center for Clinical and Basic Research -CCBR, Vejle
- France (10):
  - Institut Claude Pompidou - CMRR, Nice, Alpes Maritimes
  - CHU Rennes/Hopital Sud, Rennes, Ille Et Vilaine
  - Chu De Nancy Hop D'Adultes De Brabois, Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - CHU Saint Etienne - Hopital Nord, Saint Priest En Jarez, Pays de la Loire Region
  - CHU d'Amiens-Picardie Hopital Sud, Amiens
  - CHU de Caen Hopital Cote de Nacre, Caen
  - APHM Hôpital de la Timone, Marseille
  - Hôpital de la Pitié-Salpêtrière, Paris
  - CHU Strasbourg Hôpital de Hautepierre, Strasbourg
  - Chu de Toulouse Hopital de La Grave, Toulouse
- Germany (9):
  - Praxis Dr. Erich Scholz, Böblingen, Baden-Wurttemberg
  - ISPG - Institut für Studien zur psychischen Gesundheit, Mannheim, Baden-Wurttemberg
  - Praxis für Neurologie und Psychiatrie Dr. med. Roth, Ostfildern, Baden-Wurttemberg
  - Neurozentrum Sophienstraße, Stuttgart, Baden-Wurttemberg
  - Klinikum der Universität München, München, Bavaria
  - Klinikum Rechts der Isar der TU München, München, Bavaria
  - Neuropraxis München Süd, Unterhaching, Bavaria
  - Diakoniekrankenhaus Henriettenstiftung Hannover, Hanover, Lower Saxony
  - MVZ LiO Berlin, Berlin
- Italy (10):
  - Policlinico Univ. Agostino Gemelli, Rome, Lazio
  - Spedali Civili - Universita degli Studi, Brescia
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Ente Ospedaliero Ospedali Galliera, Genova
  - IRCCS Azienda Ospedaliera Universitaria San Martino, Genova
  - SDN - Istituto di Ricerca Diagnostica e Nucleare, Napoli
  - Azienda Ospedaliera - Universitaria Pisana, Pisa
  - IRCCS Santa Lucia, Roma
  - Universita La Sapienza, Roma
  - Azienda Ospedaliera Citta della Salute della Scienza Torino, Torino
- Japan (31):
  - Shinwakai Yachiyo Hospital, Anjo-shi, Aichi-ken
  - Nagoya Ekisaikai Hospital, Nagoya, Aichi-ken
  - Kojunkai Daido Hospital, Nagoya, Aichi-ken
  - Inage Neurology and Memory Clinic, Chiba, Chiba
  - Ehime University Hospital, Toon-Shi, Ehime
  - Takeda General Hospital, Aizu-Wakamatsu, Fukushima
  - Jisenkai Nanko Psychiatric Institute, Shirakawa-shi, Fukushima
  - Koseikai Kusatsu Hospital, Hiroshima, Hiroshima
  - NHO Hiroshima-Nishi Medical Center, Otaki-Shi, Hiroshima
  - Yokohama Hospital, Yokohama, Kanagawa
  - Koseikai Takeda Hospital, Kyoto, Kyoto
  - Uji Takeda Hospital, Uji-Shi, Kyoto
  - Nara Medical University Hospital, Kashihara, Nara
  - JADECOM Nara City Hospital, Nara, Nara
  - Oita University Hospital, Yufu-shi, Oita Prefecture
  - Katayama Medical Clinic, Kurashiki-shi, Okayama-ken
  - Himuro Neurology Clinic, Osaka, Osaka
  - Kotobukikai Tominaga Clinic, Osaka, Osaka
  - Kousaiin Hospital, Suita-shi, Osaka
  - NHO Hizen Psychiatric Center, Kanzaki-gun, Saga-ken
  - Shimizu Hospital, Shizuoka, Shizuoka
  - Memory Clinic Ochanomizu, Bunkyo-ku, Tokyo
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - Musashino Red Cross Hospital, Musashino, Tokyo
  - Keikokai P-One Clinic, Hachioji-shi, Tokyo-To
  - JOHAS Sanin Rosai Hospital, Yonago-shi, Tottori
  - Aomori Prefectural Centeral Hospital, Aomori
  - Ikeuchi Psycho Induced Internal Clinic, Kobe
  - Yuge Hospital, Kumamoto
  - NHO Niigata Hospital, Niigata
  - NHO Hokkaido Medical Center, Sapporo
- Mexico (8):
  - Hospital Universitario de Saltillo, Saltillo, Coahuila
  - Clinical Research Institute S C, Tlalnepantla, Edo de Mex
  - Mexico Centre for Clinical Research SA de CV, Mexico City, Mexico City
  - Hospital Univ. Jose Eleuterio Gonzalez, Monterrey, N.L.
  - Accelerium Clinical Research, Monterrey, Nuevo León
  - Centro de Estudios Clinicos y Esp Medicas SC, Monterrey, Nuevo León
  - Avix Investigación Clínica, S.C, Monterrey, Nuevo León
  - Instituto de Informacion en Salud Mental (INFOSAM), Monterrey, Nuevo León
- Netherlands (5):
  - Emotional Brain B.V., Almere Stad
  - Brain Research Center, Amsterdam
  - Amphia Ziekenhuis, Breda
  - EB Utrecht, Utrecht
  - Isala Klinieken, Zwolle
- Poland (12):
  - NZOZ Wroclawskie Centrum Alzheimerowskie, Wroclaw, Lower Silesian Voivodeship
  - Podlaskie Centrum Psychogeriatrii, Bialystok, Podlaskie Voivodeship
  - Uniwersyteckie Centrum Kliniczne, Gdansk, Pomeranian Voivodeship
  - NZOZ Mach-Med, Chorzów
  - Klinika Neurologii Neuro-Care, Katowice
  - Globe Badania Kliniczne SP Z O.O., Kłodzko
  - Prywatny Gabinet Lekarski U.Chyrchel, Lublin
  - Centrum Medyczne Medyk, Rzeszów
  - Euromedis Sp. z o.o., Szczecin
  - Clinsante Centrum Medyczne, Torun
  - Centrum Medyczne, Warsaw
  - Specjalistyczny Osrodek Medycyny Wieku Dojrzalego SOMED, Warsaw
- Portugal (3):
  - Hospital Fernando Fonseca, Amadora
  - Hospital de Braga, Braga
  - Hospitals da Universidade de Coimbra, Coimbra
- Russia (11):
  - SAIH Republ. Clinical Hospital of the MoH of Republ. Tatarst, Kazan'
  - SIH Kemerovo Regional Clinical Hosptial, Kemerovo
  - FSBIH Siberian Clinical Center of FMBA, Krasnoyarsk
  - LLC City Neurological Centre Sibneuromed, Novosibirsk
  - Novosibirsk State Medical University, Novosibirsk
  - Ultramed, Omsk
  - LLC Treatment and Rehabilitation, Rostov-on-Don
  - Bekhterev Psyconeurological Institute, Saint Petersburg
  - Central Medical Sanitary Hospital #122, Saint Petersburg
  - RSBIH Smolensk Regional Clinical Hospital, Smolensk
  - Regional State Institution of Healthcare Tomsk Clinica Psych, Tomsk
- South Korea (10):
  - Dong-A University Medical Center, Busan, Busan Gwang'yeogsi
  - The Catholic University of Korea-Bucheon St. Mary's Hospital, Bucheon-si, Gyeonggi-do
  - Myongji Hospital, Goyang-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Inha University Hospital, Incheon
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Hanyang University Medical Center, Seoul
  - Konkuk University Hospital, Seoul
  - Samsung Medical Center, Seoul
- Spain (9):
  - Hospital Cardiovascular San Vicente, San Vicent del Raspeig, Alicante
  - Hospital General de Catalunya, Sant Cugat del Vallès, Barcelona
  - Hospital Mutua de Terrassa, Terrassa, Barcelona
  - Hospital Virgen Del Puerto, Plasencia, Caceres
  - Policlinica Guipuzcoa, Donostia / San Sebastian, Guipuzcoa
  - Hospital Ntra Sra Perpetuo Socorro, Albacete
  - Hospital del Mar, Barcelona
  - Fundacion ACE-Institut Catala de Neurociences Aplicades, Barcelona
  - Hospital Universitario La Fe de Valencia, Valencia
- Taiwan (9):
  - Cardinal Tien Hospital, Sindian City, Taipei
  - National Taiwan University Hospital, Douliu, Yunlin County
  - Changhua Christian Hospital, Changhua
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital - Kaohsiung, Kaohsiung City
  - Taipei Medical University- Shuang Ho Hospital, New Taipei City
  - National Cheng Kung University Hospital, Tainan
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital - Linkou, Taoyuan
- United Kingdom (8):
  - Royal Devon and Exeter Hospital, Exeter, Devon
  - Re-Cognition Health Ltd, Plymouth, Devon
  - Charlton Lane Hospital, Cheltenham, Gloucestershire
  - Re-Cognition Health Ltd, Guildford, Surrey
  - Murray Royal Hospital, Perth, Tayside Region
  - Victoria Centre, Swindon, Wiltshire
  - Glasgow Memory Clinic, Glasgow
  - Re-Cognition Health Ltd, London

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://www.clinicalstudydatarequest.com/

REFERENCES:
- [Derived] Wessels AM, Tariot PN, Zimmer JA, Selzler KJ, Bragg SM, Andersen SW, Landry J, Krull JH, Downing AM, Willis BA, Shcherbinin S, Mullen J, Barker P, Schumi J, Shering C, Matthews BR, Stern RA, Vellas B, Cohen S, MacSweeney E, Boada M, Sims JR. Efficacy and Safety of Lanabecestat for Treatment of Early and Mild Alzheimer Disease: The AMARANTH and DAYBREAK-ALZ Randomized Clinical Trials. JAMA Neurol. 2020 Feb 1;77(2):199-209. doi: 10.1001/jamaneurol.2019.3988. PMID 31764959
- [Derived] Cebers G, Alexander RC, Haeberlein SB, Han D, Goldwater R, Ereshefsky L, Olsson T, Ye N, Rosen L, Russell M, Maltby J, Eketjall S, Kugler AR. AZD3293: Pharmacokinetic and Pharmacodynamic Effects in Healthy Subjects and Patients with Alzheimer's Disease. J Alzheimers Dis. 2017;55(3):1039-1053. doi: 10.3233/JAD-160701. PMID 27767991
- See also: Click here for more information about this study: A Study of LY3314814 in Participants With Mild Alzheimer's Disease Dementia (DAYBREAK-ALZ) — https://lillytrialguide.com/en/studies/mild-alzheimer's%20disease/AZET#?postal=
- See also: CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=16024&attachmentIdentifier=57afcbfd-0b6e-419e-bfa4-31474a88e3b0&fileName=CSP_NCT02783573.pdf&versionIdentifier=
- See also: SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=16024&attachmentIdentifier=88ccbed4-c60c-4494-8962-a9b57b36e8de&fileName=SAP_NCT02783573.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study consists of Placebo-Controlled Treatment Period (Weeks 0 to 78) and Delayed-Start Period (Weeks 78 to 156).
Pre-assignment Details: In Period 1, per the protocol, placebo-controlled groups (Placebo for 78 weeks then Lanabecestat 20 mg; Placebo for 78 weeks then Lanabecestat 50 mg) were combined to form one placebo group. As study terminated early and very few participants entered into the period 2, the arms in period 2 are combined based on dose exposure for ease of comparison.
Groups:
- Placebo: Participants received placebo film-coated oral tablets once daily.
- Lanabecestat 20 Milligrams (mg): Participants received lanabecestat 20 mg film-coated oral tablets once daily.
- Lanabecestat 50 mg: Participants received lanabecestat 50 mg film-coated oral tablets once daily.
Period: Placebo-Controlled Treatment Period
Arm/Group | Placebo | Lanabecestat 20 Milligrams (mg) | Lanabecestat 50 mg
Started | 562 | 590 | 570
Received at Least 1 Dose of Study Drug | 558 | 588 | 568
Completed | 26 | 28 | 22
Not Completed | 536 | 562 | 548
Not completed — Adverse Event | 13 | 17 | 13
Not completed — Death | 4 | 2 | 3
Not completed — Lack of Efficacy | 0 | 0 | 2
Not completed — Lost to Follow-up | 3 | 3 | 1
Not completed — Non-Compliance | 0 | 1 | 0
Not completed — Other-determined by Investigator | 0 | 1 | 2
Not completed — Physician Decision | 3 | 1 | 3
Not completed — Protocol Violation | 1 | 2 | 0
Not completed — Withdrawal by Subject | 15 | 20 | 23
Not completed — Withdrawal due to Caregiver Circumstance | 3 | 3 | 9
Not completed — Sponsor Decision | 494 | 512 | 492
Period: Delayed-Start Period
Arm/Group | Placebo | Lanabecestat 20 Milligrams (mg) | Lanabecestat 50 mg
Started | 0 (Participants from placebo group were randomized to Lanabecestat 20 mg and 50 mg.) | 17 (Participants completed period 1 may not have entered period 2 due to early termination of the study.) | 12 (Participants completed period 1 may not have entered period 2 due to early termination of the study.)
Received at Least 1 Dose of Study Drug | 0 | 14 | 12
Completed | 0 | 0 | 0
Not Completed | 0 | 17 | 12
Not completed — Sponsor Decision | 0 | 17 | 12

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study drug.
Groups:
- Lanabecestat 20 mg: Participants received lanabecestat 20 mg film-coated oral tablets once daily.
- Total: Total of all reporting groups
Arm/Group | Placebo | Lanabecestat 20 mg | Lanabecestat 50 mg | Total
Number analyzed (Participants) | 562 | 590 | 570 | 1722
Age, Continuous [Mean (Standard Deviation); unit: Years] | 72.1 (7.1) | 72.3 (7.0) | 72.6 (7.0) | 72.3 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 348 | 335 | 340 | 1023
  Male | 214 | 255 | 230 | 699
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 53 | 45 | 55 | 153
  Not Hispanic or Latino | 416 | 442 | 423 | 1281
  Unknown or Not Reported | 93 | 103 | 92 | 288
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 7 | 6 | 18
  Asian | 64 | 76 | 69 | 209
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 3 | 4
  Black or African American | 4 | 5 | 9 | 18
  White | 387 | 398 | 389 | 1174
  More than one race | 72 | 70 | 62 | 204
  Unknown or Not Reported | 30 | 33 | 32 | 95
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 196 | 205 | 199 | 600
  Czechia | 42 | 42 | 45 | 129
  Japan | 38 | 43 | 38 | 119
  United Kingdom | 23 | 22 | 23 | 68
  Portugal | 8 | 8 | 8 | 24
  Russia | 33 | 36 | 31 | 100
  Spain | 25 | 25 | 28 | 78
  Canada | 32 | 33 | 31 | 96
  South Korea | 19 | 20 | 20 | 59
  Netherlands | 9 | 9 | 12 | 30
  China | 1 | 0 | 1 | 2
  Taiwan | 5 | 10 | 9 | 24
  Poland | 39 | 43 | 40 | 122
  Denmark | 7 | 8 | 8 | 23
  Italy | 23 | 22 | 21 | 66
  Mexico | 11 | 9 | 9 | 29
  France | 30 | 33 | 30 | 93
  Germany | 21 | 22 | 17 | 60
ADAS-Cog13 (13-item Alzheimer's Disease Assessment Scale) [Mean (Standard Deviation); unit: Units on a Scale] — ADAS-Cog13, a 13-item rating scale, measured the severity of cognitive dysfunction in persons with Alzheimer's disease (AD). Scores ranged from 0 to 85, with a higher score indicating worse cognitive functioning.
  Units on a Scale | 30.4 (7.9) | 30.6 (8.3) | 30.6 (8.5) | 30.5 (8.2)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Alzheimer´s Disease Assessment Scale- Cognitive Subscale (ADAS-Cog13) Score
Description: ADAS-Cog13 (13-item version of ADAS Cog) is a psychometric instrument that evaluates word recall, ability to follow commands, constructional praxis, naming, ideational praxis, orientation, word recognition, memory, comprehension of spoken language, word-finding, and language ability, with a measure of delayed word recall and concentration/ distractibility. The total score of the 13-item scale ranges from 0 to 85, with an increase in score indicating cognitive worsening. Least Squares (LS) mean was determined by mixed-model repeated measures (MMRM) model with factors for treatment, visit, treatment-by-visit interaction, acetylcholinesterase Inhibitor (AChEI) use at baseline, pooled site, and covariates for baseline ADAS-Cog13 total score, age at baseline, and baseline ADAS-Cog13 total score-by-visit interaction.
Time Frame: Baseline, Week 78
Population: All randomized participants who received at least one dose of study drug and have baseline and at least one post-baseline data for ADAS-Cog13 measure.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Lanabecestat 20 mg | Lanabecestat 50 mg
Number analyzed (Participants) | 460 | 471 | 464
Units on a scale | 6.42 (1.23) | 8.93 (1.11) | 6.20 (1.32)
Statistical Analysis 1: Comparison: Placebo vs Lanabecestat 20 mg; Test type: Superiority; p = 0.129, Mixed Models Analysis; LS Mean Difference (Final Values) = 2.51, 95% CI 2-sided [-0.752 to 5.776], Standard Error of Mean 1.64
Statistical Analysis 2: Comparison: Placebo vs Lanabecestat 50 mg; Test type: Superiority; p = 0.903, Mixed Models Analysis; LS Mean Difference (Final Values) = -0.21, 95% CI 2-sided [-3.725 to 3.296], Standard Error of Mean 1.76

2. Secondary Outcome: Change From Baseline in Alzheimer´s Disease Cooperative Study Activities of Daily Living Inventory Instrumental Items Score (ADCS-iADL)
Description: The ADCS-ADL is a 23-item inventory developed as a rater-administered questionnaire answered by the participant's caregiver. The ADCS-ADL measures both basic and instrumental activities of daily living by participants. The range for the ADCS-iADL is 0-59 with higher scores reflecting better performance. LS Mean was determined by MMRM model with factors for treatment, visit, treatment-by-visit interaction, AChEI use at baseline, pooled site, and covariates for baseline iADL score, age at baseline, and baseline iADL score-by-visit interaction.
Time Frame: Baseline, Week 78
Population: All randomized participants who received at least one dose of study drug and have baseline and at least one post-baseline data for ADCS-iADL measure.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Lanabecestat 20 mg | Lanabecestat 50 mg
Number analyzed (Participants) | 357 | 369 | 347
Units on a scale | -3.95 (1.27) | -6.91 (1.29) | -7.13 (1.40)
Statistical Analysis 1: Comparison: Placebo vs Lanabecestat 20 mg; Test type: Superiority; p = 0.100, Mixed Models Analysis; LS Mean Difference (Final Values) = -2.95, 95% CI 2-sided [-6.488 to 0.580], Standard Error of Mean 1.78
Statistical Analysis 2: Comparison: Placebo vs Lanabecestat 50 mg; Test type: Superiority; p = 0.092, Mixed Models Analysis; LS Mean Difference (Final Values) = -3.18, 95% CI 2-sided [-6.876 to 0.525], Standard Error of Mean 1.86

3. Secondary Outcome: Change From Baseline in Functional Activities Questionnaire (FAQ) Score
Description: FAQ is a 10-item, caregiver-based questionnaire and was administered to the study partner who was asked to rate the participant's ability to perform a variety of activities ranging from writing checks, assembling tax records, shopping, playing games, food preparation, traveling, keeping appointments, traveling out of neighborhood, keeping track of current events and understanding media. FAQ total score was calculated by adding the scores from each of the 10 items. Each activity is rated on a scale from 0 to 3 (Never did and would have difficulty now=1; never did [the activity] but could do now=0; normal=0; has difficulty but does by self=1; requires assistance=2; Dependent =3). FAQ scale is 0 to 30, with higher scores indicating greater impairment. LS Mean determined by MMRM model with factors for treatment, visit, treatment-by-visit interaction, AChEI use at baseline, pooled site, and covariates for baseline FAQ total score, by-visit interaction and age at baseline.
Time Frame: Baseline, Week 78
Population: All randomized participants who received at least one dose of study drug and have baseline and at least one post-baseline data for FAQ score.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Lanabecestat 20 mg | Lanabecestat 50 mg
Number analyzed (Participants) | 358 | 369 | 347
Units on a scale | 3.93 (0.81) | 5.16 (0.85) | 3.41 (0.91)
Statistical Analysis 1: Comparison: Placebo vs Lanabecestat 20 mg; Test type: Superiority; p = 0.285, Mixed Models Analysis; LS Mean Difference (Final Values) = 1.23, 95% CI 2-sided [-1.045 to 3.499], Standard Error of Mean 1.14
Statistical Analysis 2: Comparison: Placebo vs Lanabecestat 50 mg; Test type: Superiority; p = 0.661, Mixed Models Analysis; LS Mean Difference (Final Values) = -0.52, 95% CI 2-sided [-2.889 to 1.843], Standard Error of Mean 1.19

4. Secondary Outcome: Change From Baseline on the Integrated Alzheimer's Disease Rating Scale (iADRS) Score
Description: The iADRS is a composite that measures both cognition and function. The iADRS comprises scores form the ADAS- Cog and the ADCS-iADL. The iADRS is calculated as a linear combination of the total scores of the ADAS-Cog13 (score range 0 to 85 with higher scores reflecting worse performance) and the ADCS-iADL (score range from 0-59 with higher scores reflecting better performance). The iADRS score ranges from 0 to 144 with higher scores indicating greater impairment. LS Mean was determined by MMRM with factors for treatment, visit, treatment-by-visit interaction, AChEI use at baseline, pooled site, and covariates for baseline iADRS13 total score, age at baseline, and baseline iADRS13 total score-by-visit interaction.
Time Frame: Baseline, Week 78
Population: All randomized participants who received at least one dose of study drug and have baseline and at least one post-baseline data for iADRS.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Lanabecestat 20 mg | Lanabecestat 50 mg
Number analyzed (Participants) | 342 | 348 | 333
Units on a scale | -10.46 (1.97) | -15.22 (1.90) | -12.43 (2.08)
Statistical Analysis 1: Comparison: Placebo vs Lanabecestat 20 mg; Test type: Superiority; p = 0.079, Mixed Models Analysis; LS Mean Difference (Final Values) = -4.77, 95% CI 2-sided [-10.103 to 0.56], Standard Error of Mean 2.69
Statistical Analysis 2: Comparison: Placebo vs Lanabecestat 50 mg; Test type: Superiority; p = 0.486, Mixed Models Analysis; LS Mean Difference (Final Values) = -1.97, 95% CI 2-sided [-7.573 to 3.62], Standard Error of Mean 2.82

5. Secondary Outcome: Change From Baseline in the Clinical Dementia Rating - Sum of Boxes (CDR-SB) Score
Description: The CDR-SB is a rater administered scale and impairment is scored in each of categories: memory, orientation, judgment and problem solving, community affairs, home and hobbies and personal care. Impairment is scored on a scale in which no dementia = 0, questionable dementia = 0.5, mild dementia = 1, moderate dementia = 2 and severe dementia = 3. The 6 individual category ratings, or "box scores", were added together to give the CDR-Sum of Boxes which ranges from 0-18, with higher scores indicating greater impairment. LS Mean was determined by MMRM methodology with factors for treatment, visit, treatment-by-visit interaction, AChEI use at baseline, pooled site, and covariates for baseline CDR-SB score, age at baseline, and baseline CDR-SB score-by-visit interaction.
Time Frame: Baseline, Week 78
Population: All randomized participants who received at least one dose of study drug and have baseline and at least one post-baseline data for CDR-SB.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Lanabecestat 20 mg | Lanabecestat 50 mg
Number analyzed (Participants) | 369 | 370 | 363
Units on a scale | 2.32 (0.42) | 2.57 (0.41) | 2.10 (0.45)
Statistical Analysis 1: Comparison: Placebo vs Lanabecestat 20 mg; Test type: Superiority; p = 0.663, Mixed Models Analysis; LS Mean Difference (Final Values) = 0.25, 95% CI 2-sided [-0.890 to 1.391], Standard Error of Mean 0.57
Statistical Analysis 2: Comparison: Placebo vs Lanabecestat 50 mg; Test type: Superiority; p = 0.717, Mixed Models Analysis; LS Mean Difference (Final Values) = -0.22, 95% CI 2-sided [-1.423 to 0.983], Standard Error of Mean 0.60

6. Secondary Outcome: Time to Progression as Measured by Loss of Clinical Dementia Rating (CDR) Global Score Stage
Description: The CDR global score is a composite score calculated using the Washington University CDR-assignment algorithm applied to the 6 individual domain box scores (Morris 1993). The memory domain is considered the primary category that drives the CDR global outcome, and all other domains are secondary. The CDR global score ranges from 0 to 3 (0 = no dementia, 0.5 = questionable dementia, 1 = mild dementia, 2 = moderate dementia, 3 = severe dementia).
Time Frame: From Loss of 1 Global Stage through Week 78
Population: All randomized participants who received at least one dose of study drug and have baseline and at least one post-baseline data for CDR global score.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo | Lanabecestat 20 mg | Lanabecestat 50 mg
Number analyzed (Participants) | 479 | 500 | 466
Days | 379 [367 to 546] | 367 [365 to 456] | 449 [365 to 491]

7. Secondary Outcome: Change From Baseline in Neuropsychiatric Inventory (NPI) Score
Description: The NPI is a questionnaire administered to caregivers that quantifies behavioral changes. Each of the 12 behavioral domains the caregiver reports as present are scored for Frequency, scale: 1 (Occasionally) to 4 (Very Frequently), and Severity, scale: 1 (Mild) to 3 (Severe). If the domain is reported by the caregiver as 'Not Affected,' that domain is scored as 0. The individual domain scores are calculated by multiplying the frequency times the severity for each domain. NPI Total Score is calculated by adding the individual domain scores together for all 12 domains, with a scores range from 0 to 144, with higher scores indicating a greater severity of neuropsychiatric disturbance. LS Mean was determined by MMRM methodology with factors for treatment, visit, treatment-by-visit interaction, AChEI use at baseline, pooled site, and covariates for baseline NPI score, age at baseline, and baseline NPI score-by-visit interaction.
Time Frame: Baseline, Week 78
Population: All randomized participants who received at least one dose of study drug and have baseline and at least one post-baseline data for NPI.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Lanabecestat 20 mg | Lanabecestat 50 mg
Number analyzed (Participants) | 351 | 363 | 342
Units on a scale | 3.45 (1.70) | 3.75 (1.84) | 0.44 (1.45)
Statistical Analysis 1: Comparison: Placebo vs Lanabecestat 20 mg; Test type: Superiority; p = 0.899, Mixed Models Analysis; LS Mean Difference (Final Values) = 0.30, 95% CI 2-sided [-4.297 to 4.889], Standard Error of Mean 2.34
Statistical Analysis 2: Comparison: Placebo vs Lanabecestat 50 mg; Test type: Superiority; p = 0.164, Mixed Models Analysis; LS Mean Difference (Final Values) = -3.01, 95% CI 2-sided [-7.267 to 1.238], Standard Error of Mean 2.16

8. Secondary Outcome: Change From Baseline on the Mini-Mental State Examination (MMSE)
Description: The MMSE is an instrument used to assess a participant's global cognitive function. The MMSE assesses orientation to time and place, immediate and delayed recall of words, attention and calculation, language (naming, comprehension and repetition), and spatial ability (copying a figure). The range for MMSE total Score is 0 to 30, with a higher score indicating better cognitive performance. LS Mean was determined by MMRM methodology with factors for treatment, visit, treatment-by-visit interaction, AChEI use at baseline, pooled site, and covariates for baseline MMSE total score, age at baseline, and baseline MMSE total score-by-visit interaction.
Time Frame: Baseline, Week 78
Population: All randomized participants who received at least one dose of study drug and have baseline and at least one post-baseline data for MMSE.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Lanabecestat 20 mg | Lanabecestat 50 mg
Number analyzed (Participants) | 476 | 495 | 477
Units on a scale | -4.16 (0.59) | -5.43 (0.58) | -4.31 (0.64)
Statistical Analysis 1: Comparison: Placebo vs Lanabecestat 20 mg; Test type: Superiority; p = 0.126, Mixed Models Analysis; LS Mean Difference (Final Values) = -1.26, 95% CI 2-sided [-2.891 to 0.362], Standard Error of Mean 0.82
Statistical Analysis 2: Comparison: Placebo vs Lanabecestat 50 mg; Test type: Superiority; p = 0.862, Mixed Models Analysis; LS Mean Difference (Final Values) = -0.15, 95% CI 2-sided [-1.867 to 1.566], Standard Error of Mean 0.86

9. Secondary Outcome: Percent Change From Baseline in Concentration of Cerebrospinal Fluid (CSF) Biomarker Amyloid Beta (Aβ)1-42
Description: Concentration of the peptide Aβ 1-42 in plasma measured by validated immunoassay. LS Mean was determined by Analysis of covariance (ANCOVA) with last observation carried forward (LOCF), terms for treatment, baseline biomarker and age at baseline.
Time Frame: Baseline, Week 71
Population: All randomized participants who received at least one dose of study drug and have baseline and at least one post-baseline data for Aβ1-42.
Measure: Least Squares Mean (Standard Error); unit: Percent change in Aβ1-42
Arm/Group | Placebo | Lanabecestat 20 mg | Lanabecestat 50 mg
Number analyzed (Participants) | 4 | 5 | 5
Percent change in Aβ1-42 | 23.68 (26.76) | -13.87 (24.30) | -17.04 (23.26)
Statistical Analysis 1: Comparison: Placebo vs Lanabecestat 20 mg; Test type: Superiority; p = 0.343, ANCOVA; LS Mean Difference (Final Values) = -37.55, 95% CI 2-sided [-122.35 to 47.26], Standard Error of Mean 37.49
Statistical Analysis 2: Comparison: Placebo vs Lanabecestat 50 mg; Test type: Superiority; p = 0.276, ANCOVA; LS Mean Difference (Final Values) = -40.72, 95% CI 2-sided [-120.17 to 38.73], Standard Error of Mean 35.12

10. Secondary Outcome: Percent Change From Baseline in Concentration of CSF Biomarker Aβ1-40
Description: Concentration of the peptide Aβ 1-40 in plasma measured by immunoassay. LS Mean was determined by ANCOVA with LOCF (last observation carried forward), terms for treatment, baseline biomarker and age at baseline.
Time Frame: Baseline, Week 71
Population: All randomized participants who received at least one dose of study drug and have baseline and at least one post-baseline data for Aβ1-40.
Measure: Least Squares Mean (Standard Error); unit: Percent change in Aβ1-40
Arm/Group | Placebo | Lanabecestat 20 mg | Lanabecestat 50 mg
Number analyzed (Participants) | 4 | 5 | 5
Percent change in Aβ1-40 | 24.52 (23.08) | -37.42 (20.76) | -9.63 (20.74)
Statistical Analysis 1: Comparison: Placebo vs Lanabecestat 20 mg; Test type: Superiority; p = 0.079, ANCOVA; LS Mean Difference (Final Values) = -61.94, 95% CI 2-sided [-132.75 to 8.87], Standard Error of Mean 31.30
Statistical Analysis 2: Comparison: Placebo vs Lanabecestat 50 mg; Test type: Superiority; p = 0.303, ANCOVA; LS Mean Difference (Final Values) = -34.15, 95% CI 2-sided [-104.88 to 36.59], Standard Error of Mean 31.27

11. Secondary Outcome: Change From Baseline in CSF Biomarker Total Tau
Description: Cerebrospinal fluid samples were collected for analysis of concentration total tau. LS Mean was determined by ANCOVA with LOCF and with factors for treatment, baseline biomarker and age at baseline.
Time Frame: Baseline, Week 71
Population: All randomized participants who received at least one dose of study drug and have baseline and at least one post-baseline data for CSF Total Tau.
Measure: Least Squares Mean (Standard Error); unit: Picogram per milliliter (pg/mL)
Arm/Group | Placebo | Lanabecestat 20 mg | Lanabecestat 50 mg
Number analyzed (Participants) | 4 | 5 | 5
Picogram per milliliter (pg/mL) | 1.84 (9.75) | 18.16 (9.77) | -11.21 (9.32)
Statistical Analysis 1: Comparison: Placebo vs Lanabecestat 20 mg; Test type: Superiority; p = 0.283, ANCOVA; LS Mean Difference (Final Values) = 16.32, 95% CI 2-sided [-16.015 to 48.659], Standard Error of Mean 14.29
Statistical Analysis 2: Comparison: Placebo vs Lanabecestat 50 mg; Test type: Superiority; p = 0.349, ANCOVA; LS Mean Difference (Final Values) = -13.05, 95% CI 2-sided [-42.929 to 16.820], Standard Error of Mean 13.21

12. Secondary Outcome: Change From Baseline in CSF Biomarker Phosphorylated Tau
Description: Cerebrospinal fluid samples are collected for analysis of concentration of phosphorylated tau. LS Mean was determined by ANCOVA with LOCF and with factors for treatment, baseline biomarker and age at baseline.
Time Frame: Baseline, Week 71
Population: All randomized participants who received at least one dose of study drug and have baseline and at least one post-baseline data for CSF Phosphorylated Tau.
Measure: Least Squares Mean (Standard Error); unit: Picogram per milliliter (pg/mL)
Arm/Group | Placebo | Lanabecestat 20 mg | Lanabecestat 50 mg
Number analyzed (Participants) | 4 | 5 | 5
Picogram per milliliter (pg/mL) | 2.22 (1.54) | 3.81 (1.49) | 0.08 (1.41)
Statistical Analysis 1: Comparison: Placebo vs Lanabecestat 20 mg; Test type: Superiority; p = 0.494, ANCOVA; LS Mean Difference (Final Values) = 1.59, 95% CI 2-sided [-3.457 to 6.640], Standard Error of Mean 2.23
Statistical Analysis 2: Comparison: Placebo vs Lanabecestat 50 mg; Test type: Superiority; p = 0.323, ANCOVA; LS Mean Difference (Final Values) = -2.13, 95% CI 2-sided [-6.743 to 2.481], Standard Error of Mean 2.04

13. Secondary Outcome: Change From Baseline in Brain Amyloid Burden Using Florbetapir Amyloid Positron Emission Tomography (PET) Scan
Description: Amyloid deposition in the brain is one of the defining neuropathologic findings of Alzheimer's disease. Florbetapir exhibits high affinity specific binding to amyloid plaques. The change from baseline was measured as average standard uptake value ratio (SUVr) in prespecified regions of interest (ROI) assessed by florbetapir amyloid PET imaging in a subset of participants. The Centiloid scale standardizes quantitative brain amyloid PET results to allow cross-tracer and cross-methodology comparisons. The Centiloid scale anchor points are 0 and 100, where 0 represents a high-certainty amyloid negative scan and 100 represents the amount of global amyloid deposition found in a typical AD scans. Florbetapir SUVr was converted to the Centiloid scale using the following conversion: Florbetapir Centiloids = 183 x SUVr - 177. LS Mean was determined by using ANCOVA methodology with terms for treatment, baseline biomarker and age at baseline.
Time Frame: Baseline, Week 78
Population: All randomized participants who received at least one dose of study drug and have baseline and at least one post-baseline data for brain amyloid burden.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Lanabecestat 20 mg | Lanabecestat 50 mg
Number analyzed (Participants) | 7 | 10 | 7
Units on a scale | -2.43 (10.47) | -0.21 (7.79) | -17.63 (9.69)
Statistical Analysis 1: Comparison: Placebo vs Lanabecestat 20 mg; Test type: Superiority; p = 0.873, ANCOVA; LS Mean Difference (Final Values) = 2.22, 95% CI 2-sided [-26.569 to 31.017], Standard Error of Mean 13.76
Statistical Analysis 2: Comparison: Placebo vs Lanabecestat 50 mg; Test type: Superiority; p = 0.337, ANCOVA; LS Mean Difference (Final Values) = -15.20, 95% CI 2-sided [-47.488 to 17.096], Standard Error of Mean 15.43

14. Secondary Outcome: Change From Baseline in Regional Cerebral Blood Flow (rCBF) Using Florbetapir Perfusion Scan
Description: Florbetapir perfusion evaluated the regional cerebral blood flow (rCBF) as a biomarker of brain function and was performed at the same time as the amyloid florbetapir PET. Cerebral perfusion, especially in temporal and parietal areas, is reduced in AD and this pattern of hypoperfusion closely mirrors the hypometabolism pattern observed using FDG PET. Annualized change is derived as change at LOCF divided by (LOCF date - baseline date) multiplied by 365. LS Mean was determined by ANCOVA with LOCF (last observation carried forward) and with factors for treatment, baseline biomarker and age at baseline.
Time Frame: Baseline, Week 78
Population: All randomized participants who received at least one dose of study drug and have baseline and at least one post-baseline data for rCBF.
Measure: Least Squares Mean (Standard Error); unit: Standard Uptake Value ratio (SUVr)
Arm/Group | Placebo | Lanabecestat 20 mg | Lanabecestat 50 mg
Number analyzed (Participants) | 82 | 65 | 66
Standard Uptake Value ratio (SUVr) | -0.03 (0.01) | -0.03 (0.01) | -0.03 (0.01)
Statistical Analysis 1: Comparison: Placebo vs Lanabecestat 20 mg; Test type: Superiority; p = 0.927, ANCOVA; LS Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-0.015 to 0.017], Standard Error of Mean 0.01
Statistical Analysis 2: Comparison: Placebo vs Lanabecestat 50 mg; Test type: Superiority; p = 0.930, ANCOVA; LS Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-0.015 to 0.017], Standard Error of Mean 0.01

15. Secondary Outcome: Change From Baseline in Whole Brain Volume
Description: Magnetic resonance imaging (MRI) was used to evaluate the effect of lanabecestat on brain atrophy/whole brain volumes. Annualized change is derived as change at LOCF divided by (LOCF date - baseline date) multiplied by 365. LS Mean was determined by ANCOVA with LOCF and with factors for treatment, baseline volumetric magnetic resonance imaging (vMRI), intracranial volume and age at baseline.
Time Frame: Baseline, Week 78
Population: All randomized participants who received at least one dose of study drug and have baseline and at least one post-baseline data for Whole Brain Volume.
Measure: Least Squares Mean (Standard Error); unit: cm^3 (cubic centimeter)
Arm/Group | Placebo | Lanabecestat 20 mg | Lanabecestat 50 mg
Number analyzed (Participants) | 221 | 215 | 214
cm^3 (cubic centimeter) | -15.76 (0.75) | -17.38 (0.75) | -18.84 (0.76)
Statistical Analysis 1: Comparison: Placebo vs Lanabecestat 20 mg; Test type: Superiority; p = 0.127, ANCOVA; LS Mean Difference (Final Values) = -1.62, 95% CI 2-sided [-3.708 to 0.464], Standard Error of Mean 1.06
Statistical Analysis 2: Comparison: Placebo vs Lanabecestat 50 mg; Test type: Superiority; p = 0.004, ANCOVA; LS Mean Difference (Final Values) = -3.08, 95% CI 2-sided [-5.172 to -0.991], Standard Error of Mean 1.06

16. Secondary Outcome: Population Pharmacokinetics (PK): Apparent Oral Clearance of Lanabecestat
Description: The apparent oral clearance of lanabecestat was estimated using a population approach. No covariate effects were assessed as part of this analysis.
Time Frame: Predose, Week 4, 7, 19, 39, 45 and Week 71 post dose
Population: All randomized participants who received at least 1 dose of study drug with evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour (L/h)
Groups:
- Lanabecestat: Participants received Lanabecestat film-coated tablets orally.
Arm/Group | Lanabecestat
Number analyzed (Participants) | 1077
Liter per hour (L/h) | 17.4 (38.8)

17. Secondary Outcome: Population PK: Central Volume of Distribution of Lanabecestat
Description: The central volume of distribution for lanabecestat was estimated using a population approach. No covariate effects were assessed as part of this analysis.
Time Frame: Predose, Week 4, 7, 19, 39, 45 and week 71 post dose
Population: All randomized participants who received at least 1 dose of study drug with evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters (L)
Arm/Group | Lanabecestat
Number analyzed (Participants) | 1077
Liters (L) | 77.8 (198)

ADVERSE EVENTS:
Time Frame: Up To 156 Weeks
Description: All randomized participants who received at least one dose of study drug. There are gender specific adverse events, only occurring in male or female participants. The number of participants exposed has been adjusted accordingly.
Groups:
- Placebo-Period 1: Participants received placebo film-coated oral tablets once daily.
- Lanabecestat 20 Mg-Period 1: Participants received lanabecestat 20 mg film-coated oral tablets once daily.
- Lanabecestat 50 Mg-Period 1: Participants received lanabecestat 50 mg film-coated oral tablets once daily.
- Lanabecestat 20 Mg-Period 2: Participants from placebo group were randomized to receive lanabecestat 20 mg film-coated oral tablets once daily.
- Lanabecestat 50 Mg-Period 2: Participants from placebo group were randomized to receive lanabecestat 50 mg film-coated oral tablets once daily.
Arm/Group | Placebo-Period 1 | Lanabecestat 20 Mg-Period 1 | Lanabecestat 50 Mg-Period 1 | Lanabecestat 20 Mg-Period 2 | Lanabecestat 50 Mg-Period 2
All-Cause Mortality (participants affected / at risk) | 5/558 | 2/588 | 3/568 | 0/14 | 0/12
Serious Adverse Events (participants affected / at risk) | 50/558 | 50/588 | 46/568 | 0/14 | 1/12
Other Adverse Events (participants affected / at risk) | 48/558 | 69/588 | 76/568 | 5/14 | 1/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo-Period 1 (N=558) | Lanabecestat 20 Mg-Period 1 (N=588) | Lanabecestat 50 Mg-Period 1 (N=568) | Lanabecestat 20 Mg-Period 2 (N=14) | Lanabecestat 50 Mg-Period 2 (N=12)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronotropic incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Trifascicular block (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal arteriovenous malformation (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peptic ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal prolapse (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling abnormal (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sudden cardiac death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis orbital (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epididymitis (Infections and infestations) | 1/211 (1) | 1/255 (1) | 0/229 (0) | 0/5 (0) | 0/7 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Liver abscess (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Orchitis (Infections and infestations) | 1/211 (1) | 0/255 (0) | 0/229 (0) | 0/5 (0) | 0/7 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Brain contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 5 (5) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heat exhaustion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pubis fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostatic specific antigen increased (Investigations) | 0/211 (0) | 1/255 (1) | 0/229 (0) | 0/5 (0) | 0/7 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ovarian cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/347 (0) | 0/333 (0) | 1/339 (1) | 0/9 (0) | 0/5 (0)
Ovarian cancer stage ii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/347 (1) | 0/333 (0) | 0/339 (0) | 0/9 (0) | 0/5 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/211 (1) | 1/255 (1) | 0/229 (0) | 0/5 (0) | 0/7 (0)
Renal oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Brain injury (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebellar haematoma (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coma (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dementia Alzheimer's type (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 3 (3) | 3 (3) | 3 (4) | 0 (0) | 0 (0)
Toxic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device malfunction (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abnormal behaviour (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute psychosis (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adjustment disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aggression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Delusion (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paranoia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stress urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo-Period 1 (N=558) | Lanabecestat 20 Mg-Period 1 (N=588) | Lanabecestat 50 Mg-Period 1 (N=568) | Lanabecestat 20 Mg-Period 2 (N=14) | Lanabecestat 50 Mg-Period 2 (N=12)
Glaucoma (Eye disorders) | 5 (5) | 4 (4) | 3 (3) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 17 (19) | 29 (35) | 29 (39) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 1 (1) | 4 (4) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 21 (34) | 32 (37) | 34 (49) | 0 (0) | 0 (0)
Blood glucose decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thyroxine decreased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 2 (2) | 4 (4) | 9 (9) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 4/211 (4) | 4/255 (4) | 3/229 (3) | 1/5 (1) | 0/7 (0)

LIMITATIONS AND CAVEATS:
An independent assessment concluded the trial was not likely to meet the primary endpoint upon completion and therefore, trial stopped for futility.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor shall review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review.

DOCUMENTS (2):
  • Study Protocol (2016-02-05): https://cdn.clinicaltrials.gov/large-docs/73/NCT02783573/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-17): https://cdn.clinicaltrials.gov/large-docs/73/NCT02783573/SAP_001.pdf